CLINICAL TRIAL: NCT00378144
Title: A Community Pharmacy Based Investigation in the Self-Medication Area Efficacy and Safety of Sinutab and Pseudoephedrine on Subjects With Nasal Congestion Accompanied by Headache in the Setting of a Common Cold
Brief Title: Efficacy and Safety of Sinutab on Subjects in the Setting of a Common Cold
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A7801002; 2006-000058-35 (EudraCT Number)
Record Dates: First submitted 2006-09-05; First posted 2006-09-19 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Common Cold; Headache; Nasal Congestion
MeSH Terms: conditions — Common Cold; Headache; Nasal Obstruction | interventions — Pseudoephedrine; Acetaminophen; acetaminophen, phenylpropanolamine, phenyltoloxamine drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Pseudoephedrine/Paracetamol
  Interventions: Drug: Pseudoephedrine/Paracetamol

INTERVENTIONS:
Drug: Pseudoephedrine/Paracetamol — Fixed oral tablet doses, 2 tablets 3 times a day for 5 days with at least 4 hours between each treatment (morning-noon-evening) and last dose not later than 2 hours before bedtime [Paracetamol (500 mg) and Pseudoephedrine (30 mg)]
  Other Names: Sinutab

SUMMARY:
The purpose of this study is to investigate the efficacy and safety for a marketed sinus allergy product, Sinutab, in the treatment of nasal congestion and headache.

DETAILED DESCRIPTION:
In response to a mandated requirement from the Belgium Medicines Agency - rising from the perforce switch of Sinutab® to a 2 active ingredients Pseudoephedrine+Paracetamol combination - we have made a commitment to demonstrate the safety and efficacy of Sinutab®.

In agreement with the Medicines Agency, an in-use Pharmacy-based study has been designed to demonstrate efficacy and safety of Sinutab® for the approved indications (symptomatic relief in the common cold).

This will be a randomized, double blind, placebo-controlled, comparative phase 4, multi-centre study in parallel groups between Sinutab and placebo. To study the drug in it's 'natural environment', community pharmacists will function as local investigators. Approximately 25 community pharmacists will be carefully selected, and only be taken into consideration if appropriate software programs are used in their pharmacy.

This implicates that the pharmacist has a medication record of his patients at his disposal which he will use to check the exclusion criteria. They will include subjects with early (≤ 48 hours) cold symptoms of blocked nose with headache. Subjects fulfilling the inclusion/exclusion criteria will be assigned to one of the two treatment groups, according to a computer-generated randomization list. A sufficient number of subjects will be randomized in the order of their enrolment, targeting at 300 evaluable subjects at the conclusion of study.

The following information will be collected every evening from subjects during 7 days: symptom assessment, compliance, adverse events and the ability to go to work or school.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or more
* reported cold symptoms beginning ≤ 48 hours prior to visit 1
* scored ≥ 2 for each of nasal congestion and headache using the Modified Jackson Subject Evaluation Scale
* willing and able to comply with scheduled visits, treatment plan, and other study procedures
* evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial

Exclusion Criteria:

* patients without an electronic medication record in the pharmacy
* history of hypersensitivity to paracetamol or pseudoephedrine or lactose
* fever more than 38.0°C (measured by pharmacist)
* women in the fertile years who do not use a hormonal contraception or an intra-uterine device
* use of concomitant drugs, medications or treatments that could interfere with the study drug
* important intercurrent medical condition based on the available medication record of the patient. (cf. exclusion criterium 1)
* history of nasal reconstructive surgery
* alcohol and/or drug abuse within a 6-month period immediately preceding the screening visit
* any medication or indication that might point to an increased risk, associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the study personnel, would make the subject inappropriate for inclusion
* participation in other clinical trials the last three months and during study participation.
* employees of the clinical research centers, sponsor, the CRO's contracted for this study, or their immediate family members

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the sum of nasal congestion and headache sign/symptom scores | 7 days

SECONDARY OUTCOMES:
Change from baseline in the mean MSC score over the treatment days. The MSC score is defined as the sum of nasal congestion, headache, sore throat, and pressure around the eyes sign/symptom scores | 7 days
Change from baseline in the mean individual sign/symptom score, including nasal congestion, headache, sore throat, and pressure around the eyes | 7 days
Number of lost days at work or school | 7 Days
Mean scores for: (a) interference with concentration; and (b) interference with sleep for days during treatment with study medication only | 7 days
Safety evaluation by adverse event recording | 7 days
Exploratory Endpoint: time to reach the first of two consecutive total Modified Jackson Subject Evaluation Scale (MJS) scores (defined as sum of 8 signs/symptoms) ≤ 1 | Up to seven days

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth A Kruse, PhD, Study Director — JJCPPW
Locations (1):
- JJCPPW Investigational Site, Wilrijk, Antwerp, Belgium